CLINICAL TRIAL: NCT04082104
Title: Assessment of Stuttering Severity in Adults and Adolescences in Conversational and Narrative Contexts
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maria Alfons Fouad, principal investigator, Assiut University
Other Study IDs: Stuttering
Record Dates: First submitted 2019-08-31; First posted 2019-09-09 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Stuttering
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Stuttering Severity Instument version 3 — Riley's Stuttering Severity Instrument is used for the objective assessment of severity and in other examinations of stuttered speech. Current versions of the instrument measures three parameters: 1) stuttering frequency; 2) duration of selected stutters; 3) observed physical concomitants.

SUMMARY:
The aim of this study is to assess stuttering severity in both narration and conversation in adults and adolescences in order to determine which situation is more stressful so that more reliable and accurate measures for diagnosis can be done. Also this study will help in determining the best line of management of stuttering.

DETAILED DESCRIPTION:
Stuttering is a speech disorder in which the flow of speech is disrupted by involuntary repetitions and prolongations of sounds, syllables, words or phrases as well as involuntary silent pauses or blocks.

In the world, approximately 1% of the adult population suffer from stuttering. Stuttering has severe impact on the overall quality of the person's life such as anxiety, stress, shame, low self-esteem and negative affectivity .It also affects his educational attainment, his attractiveness and work life as he avoids employment.

Stuttering varies in severity, frequency and duration from situation to situation. So its dynamics are best understood within discourse contexts that involve interactions with other people. Clinicians typically rely on spontaneous conversational samples for analyzing speech disfluencies. They have good validity, but the use of a more structured form of speech may allow for more efficient, reliable elicitation of stuttering related behaviours and better understanding of the nature of stuttering.

Narration offers a more structured context than conversation because storytellers must weave together information about the characters, the circumstances and actions. Also, narration often contains more complex language than conversation and put the whole responsibility on the speaker for planning and conveying the information to the listener, compared to conversation where two or more speakers co-construct the stream of topics and comments. Thus, narration places more linguistic, cognitive and communicative demands on speakers than does conversation.

A research was done on six adult participants and showed that some of them stuttered more during conversation and others stuttered more during narration.

ELIGIBILITY:
Inclusion Criteria:

1. Age :11-50
2. Gender : both sex will be included in the study
3. IQ >85
4. No previous therapy

Exclusion Criteria:

* 1. Presence of any other speech, language, physical or neuropsychatric disorders.

Ages: 11 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Stuttering adults and adolescences will be referred from the outpatient clinic of Phoniatric Unit at Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-14 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
measuring the stuttering severity index in narrative and conversational contexts by using Stuttering Severity Instrument version 3 (scale ranges from very mild to very severe) | baseline
  Using SSI-3 to evaluate stuttering in both conversational and narrative contexts

SECONDARY OUTCOMES:
Comparison between the stuttering severity indices in narrative and conversational contexts (comparing the results of the primary outcome) by using the Statistical Package for the Social Sciences | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Byrd CT, Logan KJ, Gillam RB. Speech disfluency in school-age children's conversational and narrative discourse. Lang Speech Hear Serv Sch. 2012 Apr;43(2):153-63. doi: 10.1044/0161-1461(2011/10-0068). Epub 2012 Jan 23. PMID 22269580
- [Background] Constantino CD, Leslie P, Quesal RW, Yaruss JS. A preliminary investigation of daily variability of stuttering in adults. J Commun Disord. 2016 Mar-Apr;60:39-50. doi: 10.1016/j.jcomdis.2016.02.001. Epub 2016 Feb 23. PMID 26945438